CLINICAL TRIAL: NCT00004092
Title: Randomized Phase II Study of Adriamycin/Cytoxan/Taxol (ACT) vs. Cytoxan, Thiotepa, Carboplatin (STAMP V) in Patients With High-Risk Primary Breast Cancer
Brief Title: Combination Chemotherapy in Treating Patients With High-Risk Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 98096; U01CA063265 (NIH); P30CA033572 (NIH); CHNMC-IRB-98096; CHNMC-PHII-18; NCI-H99-0038; CDR0000067305 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Results first posted 2015-08-04 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; Carboplatin; Cyclophosphamide; Doxorubicin; Paclitaxel; Thiotepa; Peripheral Blood Stem Cell Transplantation

ARMS (2):
- Arm I (ACT) (closed to accrual as of 4/6/2006) (Experimental): Patients receive doxorubicin IV over 24 hours on days -9 to -6, cyclophosphamide IV over 2 hours on day -5, and paclitaxel IV over 24 hours on day -2. PBSC are reinfused on days -2 and 0. G-CSF is administered beginning on day 0 and continuing until blood counts recover.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel; Procedure: peripheral blood stem cell transplantation
- Arm II (STAMP V) (Active Comparator): Patients receive cyclophosphamide IV, carboplatin IV, and thiotepa IV over 24 hours on days -7 to -4. PBSC are reinfused and G-CSF is administered as in arm I.
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: cyclophosphamide; Drug: thiotepa; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim — Given IV or subcutaneously
Drug: carboplatin — Given IV
  Arms: Arm II (STAMP V)
Drug: cyclophosphamide — Given IV
Drug: doxorubicin hydrochloride — Given IV
  Arms: Arm I (ACT) (closed to accrual as of 4/6/2006)
Drug: paclitaxel — Given IV
  Arms: Arm I (ACT) (closed to accrual as of 4/6/2006)
Drug: thiotepa — Given IV
  Arms: Arm II (STAMP V)
Procedure: peripheral blood stem cell transplantation — Patients receive autologous peripheral blood stem cells

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying two different regimens of combination chemotherapy and comparing them to see how well they work in treating patients with high-risk primary stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the toxic effects of doxorubicin, cyclophosphamide, and paclitaxel vs cyclophosphamide, thiotepa, and carboplatin in patients with high-risk primary breast cancer. (Arm I closed to accural as of 4/6/2006.)
* Compare the efficacies of these regimens followed by peripheral blood stem cell rescue in these patients.
* Determine the efficacy of a bisphosphonate to prevent relapse/metastasis after high-dose chemotherapy in these patients.

OUTLINE: This is a randomized study. Patients are stratified by stage of disease.

Peripheral blood stem cells (PBSC) are collected after mobilization with filgrastim (G-CSF), administered subcutaneously or IV, twice daily beginning 3 days before collection and continuing until collection is complete.

All patients receive conventional-dose adjuvant chemotherapy, probably comprising doxorubicin IV, cyclophosphamide IV, and fluorouracil IV over 1 hour on days 1, 22, 43, and 64. Patients are then randomized to receive 1 of 2 treatment arms of high-dose chemotherapy. (Arm I closed to accrual as of 4/6/2006.)

* Arm I (ACT) (closed to accrual as of 4/6/2006): Patients receive doxorubicin IV over 24 hours on days -9 to -6, cyclophosphamide IV over 2 hours on day -5, and paclitaxel IV over 24 hours on day -2. PBSC are reinfused on days -2 and 0. G-CSF is administered beginning on day 0 and continuing until blood counts recover.
* Arm II (STAMP V): Patients receive cyclophosphamide IV, carboplatin IV, and thiotepa IV over 24 hours on days -7 to -4. PBSC are reinfused and G-CSF is administered as in arm I.

Within 4-6 weeks of day 0 of high-dose chemotherapy, patients with estrogen and/or progesterone receptor positive tumors receive oral tamoxifen twice daily for 5 years. Patients are also randomized to receive a bisphosphonate comprising pamidronate IV every 4 weeks for 2 years.

Quality of life is assessed before therapy, at 30 days after high-dose chemotherapy, and at 6 and 12 months.

Patients are followed every 3 months for 1 year and then every 6 months for at least 10 years.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven high-risk primary breast cancer with less than 60% chance of progression-free survival of 3 years from diagnosis

  * Stage II with at least 10 positive axillary nodes OR
  * Stage IIIA or IIIB
* No histologically proven bone marrow metastasis
* No CNS metastasis
* Hormone receptor status:

  * Hormone receptor status known

PATIENT CHARACTERISTICS:

Age:

* Physiological age 60 or under

Menopausal status:

* Not specified

Performance status:

* Karnofsky 80-100%

Life expectancy:

* See Disease Characteristics

Hematopoietic:

* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT or SGPT no greater than 2 times upper limit of normal
* Hepatitis B antigen negative

Renal:

* Creatinine no greater than 1.2 mg/dL
* Creatinine clearance at least 70 mL/min
* No prior hemorrhagic cystitis

Cardiovascular:

* Ejection fraction at least 55% by MUGA
* No prior significant valvular heart disease or arrhythmia

Pulmonary:

* FEV_1 at least 60% of predicted
* pO_2 at least 85 mm Hg on room air
* pCO_2 at least 43 mm Hg on room air
* DLCO at least 60% lower limit of predicted

Other:

* No other prior malignancy except squamous cell or basal cell skin cancer or stage I or carcinoma in situ of the cervix
* No CNS dysfunction that would preclude compliance
* HIV negative
* No sensitivity to E. coli-derived products
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy
* No prior doxorubicin of total dose exceeding 240 mg/m^2
* No prior paclitaxel of total dose of at least 750 mg/m^2
* No more than 12 months since prior conventional-dose adjuvant chemotherapy

Endocrine therapy:

* At least 4 weeks since prior hormonal therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No prior radiation to the left chest wall

Surgery:

* Not specified

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 1999-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Somlo, MD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (ACT): Patients receive 41.25 mg/m2 of doxorubicin IV over 24 hours on days -9 to -6, 100 mg/kg of cyclophosphamide IV over 2 hours on day -5, and 725 mg/m2 of paclitaxel IV over 24 hours on day -4. PBSC are reinfused on days -2 and 0. G-CSF at 5 ug/kg IV is administered beginning on day 0 and continuing until blood counts recover.
  filgrastim: Given IV or subcutaneously
  cyclophosphamide: Given IV
  doxorubicin hydrochloride: Given IV
  paclitaxel: Given IV
  peripheral blood stem cell transplantation: Patients receive autologous peripheral blood stem cells
- Arm II (STAMP V): Patients receive cyclophosphamide 1.5 g/m2/day IV, carboplatin 200 mg/m2/day IV, and thiotepa 125 mg/m2/day IV over 24 hours on days -7 to -4. PBSC are reinfused on day -2 and 0 and G-CSF at 5ug/kg IV is administered as in arm I.
  filgrastim: Given IV or subcutaneously
  carboplatin: Given IV
  cyclophosphamide: Given IV
  thiotepa: Given IV
  peripheral blood stem cell transplantation: Patients receive autologous peripheral blood stem cells
Period: Overall Study
Arm/Group | Arm I (ACT) | Arm II (STAMP V)
Started | 21 | 51
Completed | 21 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (ACT) | Arm II (STAMP V) | Total
Number analyzed (Participants) | 21 | 51 | 72
Age, Continuous [Median (Full Range); unit: years] | 42 [29 to 56] | 51 [28 to 61] | 50 [28 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 51 | 72
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 51 | 72

OUTCOME MEASURES:

1. Primary Outcome: Five-Year Relapse-free Survival
Description: RFS events included death or disease recurrence. Patients who did not experience disease recurrence or death were censored at the date of last follow-up. Survival rates were estimates using the Kaplan-Meier method.
Time Frame: Five years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (ACT) | Arm II (STAMP V)
Number analyzed (Participants) | 21 | 51
percentage of participants | 47 [24 to 67] | 55 [41 to 68]

2. Secondary Outcome: Five-Year Overall Survival
Description: Patients who were still alive were censored at the date of last follow-up. Survival rates were estimates using the Kaplan-Meier method.
Time Frame: Five Years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (ACT) | Arm II (STAMP V)
Number analyzed (Participants) | 21 | 51
percentage of participants | 63 [38 to 80] | 75 [60 to 84]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 8 years.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Arm I (ACT) | Arm II (STAMP V)
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/51
Other Adverse Events (participants affected / at risk) | 21/21 | 50/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (ACT) (N=21) | Arm II (STAMP V) (N=51)
Diarrhea associated with graft versus host disease (GVHD) for BMT studies (Gastrointestinal disorders) | 19 (19) | 24 (24)
Haematemesis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Leukocytes (total WBC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 21 (21) | 49 (49)
Platelets for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 21 (21) | 48 (49)
Rash/dermatitis associated with high-dose chemotherapy or BMT studies. (Skin and subcutaneous tissue disorders) | 1 (1) | 15 (15)
Rash/desquamation associated with graft versus host disease (GVHD) for BMT studies (Skin and subcutaneous tissue disorders) | 11 (11) | 17 (17)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT studies, if specified in the protocol. (Gastrointestinal disorders) | 19 (19) | 37 (37)
Transfusion: Platelets for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 20 (20) | 44 (44)
Transfusion: pRBCs for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 20 (20) | 44 (44)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 19 (19) | 27 (27)
Haemorrhage NOS (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 21 (21) | 49 (49)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 7 (7) | 7 (7)
Lymphangiopathy NOS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 10 (10) | 7 (7)
Myocardial ischemia (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 6 (6) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 13 (13) | 18 (18)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 9 (9) | 8 (8)
Conjunctival disorder (Eye disorders) | 0 (0) | 2 (2)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (1) | 1 (1)
Eye disorder (Eye disorders) | 1 (1) | 2 (2)
Vision blurred (Eye disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 28 (28)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (7) | 20 (20)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 18 (18)
Diarrhea (Somlo COH) (Gastrointestinal disorders) | 0 (0) | 19 (19)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 15 (15)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia, esophagitis, odynophagia (Somlo COH) (Gastrointestinal disorders) | 19 (19) | 8 (8)
Esophagitis (Gastrointestinal disorders) | 19 (19) | 9 (9)
Flatulence (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 15 (23)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 4 (4)
Incontinence NOS (Gastrointestinal disorders) | 1 (1) | 2 (2)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 20 (20) | 49 (49)
Nausea (Somlo COH) (Gastrointestinal disorders) | 0 (0) | 22 (22)
Proctitis (Gastrointestinal disorders) | 0 (0) | 4 (5)
Rectal pain (Gastrointestinal disorders) | 2 (2) | 5 (5)
Stomatitis/phayngitis (Somlo COH) (Gastrointestinal disorders) | 20 (20) | 32 (32)
Vomiting (Gastrointestinal disorders) | 21 (21) | 48 (48)
Vomiting (Somlo COH) (Gastrointestinal disorders) | 0 (0) | 22 (22)
Chest pain (General disorders) | 2 (2) | 5 (5)
Chills (General disorders) | 14 (14) | 22 (22)
Edema (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 18 (18) | 48 (48)
Fever (General disorders) | 1 (1) | 11 (11)
General symptom (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 11 (11)
Oedema NOS (General disorders) | 14 (15) | 27 (27)
Pain (General disorders) | 13 (19) | 23 (39)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Immune system disorder (Immune system disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 2 (2) | 3 (4)
Infection (Infections and infestations) | 0 (0) | 1 (2)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (Infections and infestations) | 1 (1) | 7 (7)
Infection NOS (Infections and infestations) | 2 (2) | 3 (3)
Infection, Bacterial (COH) (Infections and infestations) | 0 (0) | 2 (2)
Infection, Fungal (COH) (Infections and infestations) | 0 (0) | 1 (1)
Infection, Viral (COH) (Infections and infestations) | 0 (0) | 3 (3)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ADH abnormal (Investigations) | 0 (0) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 13 (13) | 18 (18)
Alanine aminotransferase increased (Investigations) | 15 (15) | 24 (24)
Alk Phos (Somlo COH) (Investigations) | 0 (0) | 8 (8)
Alkaline phosphatase increased (Investigations) | 13 (13) | 9 (9)
Aspartate aminotransferase increased (Investigations) | 13 (13) | 19 (19)
Creatinine increased (Investigations) | 0 (0) | 2 (2)
Electrocardiogram QTc interval prolonged (Investigations) | 1 (1) | 0 (0)
Hyperbilirubinemia (Investigations) | 1 (1) | 2 (2)
Hypercholesterolemia (Investigations) | 17 (17) | 12 (12)
INR increased (Investigations) | 16 (16) | 35 (35)
Leukocyte count decreased (Investigations) | 0 (0) | 1 (1)
Lymphopenia (Investigations) | 13 (13) | 39 (39)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Neutrophils (ANC) (Somlo COH) (Investigations) | 19 (19) | 46 (46)
Neutrophils/granulocytes (ANC/AGC) for BMT studies, if specified in the protocol. (Investigations) | 21 (21) | 46 (46)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Platelets (Somlo COH) (Investigations) | 19 (19) | 46 (46)
SGOT (Somlo COH) (Investigations) | 0 (0) | 10 (10)
SGPT (Somlo COH) (Investigations) | 0 (0) | 12 (12)
Serum cholesterol increased (Investigations) | 0 (0) | 1 (1)
Weight gain (Investigations) | 6 (6) | 17 (17)
Weight loss (Investigations) | 7 (7) | 13 (13)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 19 (19) | 47 (47)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 18 (18) | 45 (45)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 7 (7)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (10) | 40 (40)
Hypocalcemia (Metabolism and nutrition disorders) | 21 (21) | 45 (45)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 21 (21) | 30 (30)
Hypomagnesemia (Metabolism and nutrition disorders) | 11 (11) | 12 (12)
Hyponatremia (Metabolism and nutrition disorders) | 20 (20) | 34 (34)
Hypophosphatemia (Metabolism and nutrition disorders) | 17 (17) | 43 (43)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 10 (10)
Joint pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 9 (9)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Depressed level of consciousness (Nervous system disorders) | 4 (4) | 4 (4)
Dizziness (Nervous system disorders) | 7 (7) | 16 (16)
Extrapyramidal disorder (Nervous system disorders) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 14 (14) | 32 (32)
Neuralgia (Nervous system disorders) | 8 (9) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 3 (3) | 4 (4)
Olfactory nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 7 (7) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 17 (17) | 6 (7)
Pyramidal tract syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Taste alteration (Nervous system disorders) | 6 (6) | 12 (12)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 15 (15) | 23 (24)
Confusion (Psychiatric disorders) | 6 (6) | 4 (4)
Depression (Psychiatric disorders) | 6 (6) | 17 (17)
Euphoria (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination NOS (Psychiatric disorders) | 5 (5) | 2 (2)
Insomnia (Psychiatric disorders) | 7 (7) | 27 (27)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 4 (4)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Blood urine present (Renal and urinary disorders) | 3 (3) | 9 (9)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 2 (2) | 3 (4)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 12 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (9)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 11 (11)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 11 (14)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 16 (16) | 19 (19)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (11) | 8 (8)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 11 (15) | 18 (20)
Sweating (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 6 (6) | 13 (13)
Hemorrhage (Vascular disorders) | 1 (1) | 4 (4)
Hot flashes (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 5 (5)
Hypotension (Vascular disorders) | 14 (14) | 26 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes